## **Title of study:**

Effect of materials of vaginal ring pessary for pelvic organ prolapse on the effects of complications and patients' satisfaction: A Randomized Control Trial

**Date of document: 11th October: 2024** 

## <u>Urogynaecology Team, Princess Margaret Hospital</u>

Study on Effect of materials of vaginal ring pessary for pelvic organ prolapse on the effects of complications and patient's satisfaction: A randomized control trial Informed consent form

I hereby consent to participate in this study. I have carefully read the study participation information page. The researcher has explained the details of the study to me in detail. I understand all the benefits and risks of this study. I had the opportunity to ask questions to the researcher, and he/she answered my questions satisfactorily.

I have obtained sufficient information for this study.

If I suffer from any physical discomfort or emotional fluctuations due to my participation in this study, the researcher will treat me or refer me to treatment. I do not waive any legal rights by signing this consent form.

I understand that study participants will have access to my medical records. I also authorize these persons to access my medical records.

I understand that my identity will be kept confidential. I also allow the Clinical Research Ethics Committee and relevant statutory bodies to directly access my research data to verify the relevant clinical research data as permitted by appropriate regulations and laws and without invading my privacy.

| Date: | • | C | | | | |
|--------|----------|----------|------------|----------|------------|--------|
| Resear | cher's 1 | name (pi | rinted): l | Research | er's signa | ature: |

Participant's signature: